CLINICAL TRIAL: NCT06877741
Title: Comparative Effects of Heavy Slow Resistance Training and Eccentric Overload Training on Pain, Range of Motion, and Lower Extremity Functions in Runners With Patellar Tendinopathy
Brief Title: Comparative Effects of Heavy Slow Resistance Training and Eccentric Overload Training in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0417
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Sports Physical Therapy
Keywords: Exercise; Heavy slow resistance; Jumper's knee; Pain; Patellar tendinopathy
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Heavy Slow Resistance exercises) (Experimental)
  Interventions: Other: Group A (Heavy Slow Resistance exercises)
- Group B (Eccentric exercises). (Experimental)
  Interventions: Other: : Group B (Eccentric exercises)

INTERVENTIONS:
Other: Group A (Heavy Slow Resistance exercises) — Pre - assessment will be taken. Heavy slow resistance exercises will be given to group A and exercises of 4 sets of 10-20 repetitions will be given
  Arms: Group A (Heavy Slow Resistance exercises)
Other: : Group B (Eccentric exercises) — Sessions should be conducted 2 times per week, similar to Group A, in 3 sets of 10-20 repetitions. Exercises focus solely on eccentric loading, such as eccentric squats, eccentric leg presses, and step-down exercises.
  Arms: Group B (Eccentric exercises).

SUMMARY:
Patellar Tendinopathy (PT) also known as Jumper's knee, is characterized by multifaceted activity-related pathology causing anterior knee pain and patellar-tendon dysfunction. It most commonly affects athletic activities that involve jumping and running. Tendinopathy is most likely to be related to mechanical loading and overuse. Athletes suffer from insidious well-localized pain, typically as the athlete starts the activity. Conservative treatment is the first line of treatment in tendinopathy, however, there is no consensus regarding the best treatment. In acute conditions, relative rest rather than immobilization is preferred. The most popular non-operative treatment involves eccentric exercise (EE). It is commonly accepted that surgical treatment must be indicated in motivated patients if carefully followed conservative treatment (physical training, injections, ESWT) is unsuccessful after 3-6 months. In recent studies, isometric and heavy slow resistance (HSR) exercises have demonstrated potential for pain reduction and functional improvement in patellar tendinopathy.

A randomized controlled trial will be conducted at the Pakistan Sports Board (PSB) Coaching Center, Lahore. 18 Subjects will be randomized into two groups; Heavy slow resistance exercises plus eccentric exercises will be given to group A and exercises of 4 sets of 10-20 repetitions will be given. Group B will give Eccentric exercises in 3 sets of 10-20 repetitions. Pre-assessments will be taken through the Numeric Pain Rating Scale (NPRS) for pain, a goniometer for range of motion, Lower extremity function assessment scale to evaluate lower limb functional impairments, and a Visa-P scale for patellar dysfunction. Assessment will be done at baseline and post 4 weeks of training. Data will be analyzed using SPSS software version 21. The normality of data will be checked, and tests will be applied according to the normality of the data, either parametric or non-parametric tests will be used (within a group or between two groups).

DETAILED DESCRIPTION:
The objective of the study is to compare the effects of heavy slow resistance training and eccentric overload training on pain, range of motion, and lower extremity functions in runners with patellar tendinopathy.

.

ELIGIBILITY:
Inclusion Criteria:

* anterior knee pain located on the inferior pole of the patella for at least 3 months while practicing sport;
* age between 18 and 45 years old;
* practicing any kind of sports at least 3 times a week
* score less than 80 on the Victorian Institute of Sport Assessment-Patellar questionnaire (VISA-p).

Exclusion Criteria:

* Knee surgery within the previous 6 months;
* Chronic joint diseases;
* Corticosteroid injection in the patellar tendon within the previous 3 months;
* Anti-inflammatory, analgesic, or antibiotic medications within the previous 48 hours;
* Any other concomitant treatment for PT

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment-Patella (VISA-P) questionnaire | 4 weeks
  This brief questionnaire assesses (i) symptoms, (ii) simple tests of function and (in') ability to play sport. Six of the eight questions are scored on a visual analogue scale from 0-10 with 10 representing optimal health. The maximal VISA score for an asymptomatic, fully performing individual is 100 points and the theoretical minimum is 0 points. We found the VISA scale to have excellent short-term test retest, and inter-tester reliability both, r>0.95 as well as good short-term stability (r=0.87).(14)
NPRS | 4 weeks
  For the NPRS, the intraclass correlation coefficient (ICC) for all subjects is .76 (p < .0001). The ICC, however, is .90 (p < .0001)(15)
Goniometer | 4 weeks
  Goniometric measurements are used to quantify baseline limitations of motion, decide on appropriate therapeutic interventions, and document the effectiveness of these interventions
LEFS | 4 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. Internal consistency is α=.96 (N=107). Test-retest reliability estimates were R=.86 (95% lower limit CI=.80) for the entire sample (n=98) and R=.94 (95% lower limit CI=.89) for the subset of patients with more chronic conditions (n=31)

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board Coaching Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muaidi QI. Rehabilitation of patellar tendinopathy. J Musculoskelet Neuronal Interact. 2020 Dec 1;20(4):535-540. PMID 33265081
- [Background] Lee WC, Ng GY, Zhang ZJ, Malliaras P, Masci L, Fu SN. Changes on Tendon Stiffness and Clinical Outcomes in Athletes Are Associated With Patellar Tendinopathy After Eccentric Exercise. Clin J Sport Med. 2020 Jan;30(1):25-32. doi: 10.1097/JSM.0000000000000562. PMID 31855909
- [Background] Schwartz A, Watson JN, Hutchinson MR. Patellar Tendinopathy. Sports Health. 2015 Sep-Oct;7(5):415-20. doi: 10.1177/1941738114568775. Epub 2015 Jan 23. PMID 26502416
- [Background] Rudavsky A, Cook J. Physiotherapy management of patellar tendinopathy (jumper's knee). J Physiother. 2014 Sep;60(3):122-9. doi: 10.1016/j.jphys.2014.06.022. Epub 2014 Aug 3. No abstract available. PMID 25092419
- [Background] Visnes H, Bahr R. The evolution of eccentric training as treatment for patellar tendinopathy (jumper's knee): a critical review of exercise programmes. Br J Sports Med. 2007 Apr;41(4):217-23. doi: 10.1136/bjsm.2006.032417. Epub 2007 Jan 29. PMID 17261559
- [Background] Rodriguez-Merchan EC. The treatment of patellar tendinopathy. J Orthop Traumatol. 2013 Jun;14(2):77-81. doi: 10.1007/s10195-012-0220-0. Epub 2012 Dec 28. PMID 23271268
- [Background] van Rijn D, van den Akker-Scheek I, Steunebrink M, Diercks RL, Zwerver J, van der Worp H. Comparison of the Effect of 5 Different Treatment Options for Managing Patellar Tendinopathy: A Secondary Analysis. Clin J Sport Med. 2019 May;29(3):181-187. doi: 10.1097/JSM.0000000000000520. PMID 31033610
- [Background] Lin PC, Hsu WY, Lee PY, Hsu SH, Chiou SS. Insights into Hepatocellular Carcinoma in Patients with Thalassemia: From Pathophysiology to Novel Therapies. Int J Mol Sci. 2023 Aug 10;24(16):12654. doi: 10.3390/ijms241612654. PMID 37628834
- [Background] Ghosh S, Cotta KB, Hande AA, Fernandes M, Mehra S. PNA-mediated efflux inhibition as a therapeutic strategy towards overcoming drug resistance in Mycobacterium smegmatis. Microb Pathog. 2021 Feb;151:104737. doi: 10.1016/j.micpath.2021.104737. Epub 2021 Jan 13. PMID 33453316
- [Background] Chung H, Lee S, Kim GA, Kim WH. Down-expression of klotho in canine mammary gland tumors and its prognostic significance. PLoS One. 2022 Jun 6;17(6):e0265248. doi: 10.1371/journal.pone.0265248. eCollection 2022. PMID 35666743
- [Background] Caradu C, Dubourg AP, Colacchio EC, Midy D, Berard X, Ducasse E. Endovascular Treatment of Complex Aneurysms with the Use of Covera Stent Grafts. J Vasc Interv Radiol. 2019 Dec;30(12):1942-1948.e1. doi: 10.1016/j.jvir.2019.05.004. Epub 2019 Sep 14. PMID 31530494
- [Background] Shen J, Li X, Yan X. Mechanical and Acoustic Properties of Jute Fiber-Reinforced Polypropylene Composites. ACS Omega. 2021 Nov 13;6(46):31154-31160. doi: 10.1021/acsomega.1c04605. eCollection 2021 Nov 23. PMID 34841157
- [Background] Martindale S, Mableson H, Bodimeade C, Hume H, Badia X, Karim J, Mahmood ASMS, Chiphwanya J, Rimal P, Boko-Collins P, Bougma R, Agyemang D, Alomatu B, Cisse A, Bathiri SA, Shu'aibu J, Betts H, Kelly-Hope LA, Riches N. The development and roll-out of a new hydrocoele surgery facility assessment tool for the elimination of lymphatic filariasis. Int Health. 2022 Sep 21;14(Suppl 2):ii55-ii63. doi: 10.1093/inthealth/ihac020. PMID 36130253
- [Background] Visentini PJ, Khan KM, Cook JL, Kiss ZS, Harcourt PR, Wark JD. The VISA score: an index of severity of symptoms in patients with jumper's knee (patellar tendinosis). Victorian Institute of Sport Tendon Study Group. J Sci Med Sport. 1998 Jan;1(1):22-8. doi: 10.1016/s1440-2440(98)80005-4. PMID 9732118
- [Background] Pearce L. Recovery through suggestion. Nurs Stand. 2013 Jul 3-9;27(44):20. doi: 10.7748/ns2013.07.27.44.20.s28. PMID 23940935
- [Background] Jacobs K. Marketing occupational therapy. Am J Occup Ther. 1987 May;41(5):315-20. doi: 10.5014/ajot.41.5.315. PMID 3688145
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543